CLINICAL TRIAL: NCT00486408
Title: A Phase 1B Open-label Clinical Trial to Expand the Characterization of the Immune Responses to the Merck Adenovirus Serotype 5 HIV-1 Gag/Pol/Nef Vaccine in Healthy, HIV-1-uninfected Adult Participants
Brief Title: Expanded Characterization of Immune Response to Merck Adenovirus 5 Gag/Pol/Nef Vaccine Given to HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 071; 10503 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; Adenovirus
MeSH Terms: conditions — HIV Infections; Adenoviridae Infections

ARMS (1):
- 1 (Experimental): MRKAd5 HIV-1 gag/pol/nef vaccine administered as 1 ml in either deltoid at study entry and Weeks 4 and 26
  Interventions: Biological: MRKAd5 HIV-1 gag/pol/nef

INTERVENTIONS:
Biological: MRKAd5 HIV-1 gag/pol/nef — 1.5x10^10 Ad vg

SUMMARY:
The purpose of this study is to intensively characterize the immune response, particularly the T-cell response, to a three-dose regimen of an adenovirus-based HIV-1 vaccine in HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will look for relationships among the immune responses induced by MRKAd5 HIV-1 gag/pol/nef vaccine. The study will also determine if the T cells that respond to different vaccine epitopes have correspondingly different functional profiles. The study will evaluate the safety and tolerability of the vaccine regimen as well.

This study will last 60 weeks. All enrolled participants will receive vaccinations at Weeks 0, 4, and 26. There will be between 8 and 20 study visits including the screening visit, depending on the site location. A physical exam, interview, and blood collection will occur at most or all visits. All participants will undergo leukapheresis approximately 4 weeks after their last vaccination and at Week 52. Medical history, an HIV test, a pregnancy test, and HIV and risk reduction counseling will occur at selected visits. Additional blood collection is now occurring in this study to collect more information about the relationship between the immune response and efficacy to the vaccine.

ELIGIBILITY:
Note: As of 09/19/07, enrollment and vaccinations have been discontinued.

Inclusion Criteria:

* Good general health
* HIV uninfected
* Weight of 110 pounds or greater
* Have access to a participating HIV Vaccine Trials Unit (HVTU) and are willing to be followed during the study
* Willing to receive HIV test results
* Understand the vaccination procedure
* Willing to use acceptable methods of contraception for at least 21 days prior to study entry and until the last study visit

Exclusion Criteria:

* HIV vaccines or placebos in prior HIV trial. Participants who can provide documentation that they received a placebo in a prior HIV trial may be eligible.
* Immunosuppressive medications within 168 days prior to first study vaccination
* Blood products within 90 days prior to first study vaccination or within 14 days after the injection
* Immunoglobulin within 90 days prior to first study vaccination or within 14 days after the injection
* Live attenuated vaccines within 42 days prior to first study vaccination or within 14 days after the injection
* Investigational research agents within 30 days prior to first study vaccination
* Medically indicated subunit or killed vaccines within 5 days prior to first study vaccination or within 14 days after the injection
* Allergy treatment with antigen injections within 30 days prior to first study vaccination
* Clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health
* Any medical, psychiatric, or social condition that, in the opinion of the investigator, would interfere with the study.
* History of anaphylaxis and/or allergy to vaccine components
* Autoimmune disease or immunodeficiency
* Uncontrolled hypertension
* Bleeding disorder
* Cancer. Participants with surgically removed cancer that is unlikely to recur are not excluded.
* Seizure disorder
* Absence of the spleen
* Abnormal laboratory values
* Mental illness that would interfere with the study
* Hysterectomy
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Relatedness of different immune response to vaccine | Throughout study
Features and number of HIV-specific CD4 and CD8 T cells produced in response to the vaccine | Throughout study
Characterization of different functions of T cells that have responded to the vaccine | Throughout study
Safety and tolerability of three doses of vaccine | Throughout study

SECONDARY OUTCOMES:
Changes in physical features of certain immune cells in response to the vaccine | Throughout study
Indications of an immune response to the vaccine | Throughout study
Presence of T cells in the genital tract | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ann Duerr, MD, PhD, MPH, Study Chair — HVTN Core Operations Center, Fred Hutchinson Cancer Research Center (FHCRC); Mike Keefer, MD, Study Chair — University of Rochester
Locations (4):
- United States (4):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Background] Barouch DH, Nabel GJ. Adenovirus vector-based vaccines for human immunodeficiency virus type 1. Hum Gene Ther. 2005 Feb;16(2):149-56. doi: 10.1089/hum.2005.16.149. PMID 15761255
- [Background] Horton H, Russell N, Moore E, Frank I, Baydo R, Havenar-Daughton C, Lee D, Deers M, Hudgens M, Weinhold K, McElrath MJ. Correlation between interferon- gamma secretion and cytotoxicity, in virus-specific memory T cells. J Infect Dis. 2004 Nov 1;190(9):1692-6. doi: 10.1086/424490. Epub 2004 Sep 30. PMID 15478077
- [Background] Tobery TW, Dubey SA, Anderson K, Freed DC, Cox KS, Lin J, Prokop MT, Sykes KJ, Mogg R, Mehrotra DV, Fu TM, Casimiro DR, Shiver JW. A comparison of standard immunogenicity assays for monitoring HIV type 1 gag-specific T cell responses in Ad5 HIV Type 1 gag vaccinated human subjects. AIDS Res Hum Retroviruses. 2006 Nov;22(11):1081-90. doi: 10.1089/aid.2006.22.1081. PMID 17147493